CLINICAL TRIAL: NCT02541552
Title: Effect of Volume of Local Anesthetic for Adductor Canal Block on Quadriceps Muscle Function: A Dose Finding Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Rakesh Sondekoppam Vijayashankar, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ADDCAN05
Record Dates: First submitted 2015-03-17; First posted 2015-09-04 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Postoperative Pain
Keywords: Knee arthroscopy; Quadriceps weakness; ropivacaine; saphenous nerve block; Adductor canal
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Knee arthroscopic patient (Experimental): 1) Male and females 2) Age 16-60 years 3) Scheduled surgery 4) Knee arthroscopy 5) ASA Class I - III
  Volume finding study to follow up-and-down design using a single cohort of patients. Intervention of patient will be dependent on effect of previous patients dose of and response to Ropivacaine 0.5% injectate.
  Interventions: Drug: Ropivacaine 0.5%

INTERVENTIONS:
Drug: Ropivacaine 0.5% — Varying volume according to motor response of previous subject
  Other Names: Naropin

SUMMARY:
Adductor canal block is commonly offered to provide pain relief following knee surgery with the hope that they cause less leg weakness than traditionally performed femoral nerve block. Infrequently, adductor canal blocks also result in leg weakness thereby potentially limiting the advantages of the technique. Investigators want to find out the effective dose for a 30% response (volume of local anesthetic which would result in clinically significant weakness of the leg)

DETAILED DESCRIPTION:
This is a sequential design method of binary response variables for determination of the dose associated with the 50% point along the dose-response curve required to cause quadriceps weakness following adductor canal bock for knee arthroscopic procedures. It is a Dixon and Massey up-and-down study design.

The primary objective is finding the EV50 of 0.5% ropivacaine needed to cause a 30% reduction in quadriceps function 20 minutes post-procedure.

This study design was selected to allow the estimation of the target dose associated with the given outcome of quadriceps weakness. The study will be performed on 36 patients undergoing knee arthroscopic procedures. The quadriceps strength on both legs will be evaluated preoperatively by the physiotherapist.

The quadriceps function will be measured using a hand held dynamometer (HDD). For quadriceps muscle strength evaluation, investigators will place the patient in a seated position with the knees flexed 60 degrees. To avoid interrater reliability (when the strength of the subject overcomes the strength of the tester) investigators will fix the HHD for quadriceps evaluation. A non-elastic strap with Velcro closures will be used to fix the HHD. The Velcro strap will be attached to a chair leg and around the subject's ankle, perpendicular to the lower leg. The HHD will be placed under the Velcro strap, on the anterior surface of the tibia, 5 cm above the transmalleolar axis.

Subjects will be educated about the procedure before outcome assessments. They will be instructed to take 2 seconds to reach maximum effort, maintain this force for 3 seconds, and then relax. For each assessment, the subjects will perform 3 consecutive contractions, separated by a 30-second pause between each trial. Investigators will use the mean value at each time point for calculations, and calculated muscle strength as percent of baseline value. An independent investigator not involved in the performance of the block will assess the quadriceps muscle function before, 20 minutes and then 4 hours after the block.

Following initial motor assessment the patients will be taken to the block room for the blocks to be performed using standard monitors which will include NIBP and pulse oximetry.

Patients will be sedated with fentanyl and midazolam titrated to effect and supplemental oxygen will be administered.The first patient will be given 30ml of ropivacaine 0.5% in the adductor canal block.

Depending on post-operative quadriceps function, the dose for the subsequent patient will either be increased by 2ml or decreased by 2ml (of the same concentration).

The adductor canal block procedure will be standardised for each patients. All patients will receive ultrasound guided saphenous nerve block in the adductor canal using 0.5% ropivacaine. After preparing the skin with chlorhexidine in alcohol solution and draping the area, the puncture sites will be infiltrated with 2% lidocaine. A 22 gauge 90 mm peripheral nerve stimulation block needle will be introduced deep to the sartorius muscle using ultrasonography and a linear high frequency probe and 30 ml (initially) of 0.5% ropivacaine will be injected after negative aspiration for blood while observing the spread of injectate.

The injection will be done above the level where the descending genicular artery is taking off from the femoral artery. The cutaneous analgesia over the medial aspect of leg will be tested to evaluate the success of saphenous nerve block 20 minutes after injection. If the descending genicular artery is not visualised on ultrasound, then the block will be performed proximal to where the femoral artery enters the hiatus in adductor magnus.

Total duration of performance and the time for the onset of sensory block in saphenous distribution will be recorded after the performance of the block. The failure rate of saphenous nerve block will be determined by the performer. Patients with failure of saphenous nerve block will be excluded from the efficacy part of the study.

After performance of the blocks, the patient will be moved to the operating room for the surgery under general anesthesia according to the choice of the anesthesiologist.

The patients will be assessed for the severity of pain after arrival in the PACU for four hours. Patients quadriceps function will be measured at 4 hours post-operatively. Complications such as bruising and post-block neurological deficits will be prospectively collected.

ELIGIBILITY:
Inclusion Criteria:

* Male and females
* Age 16-60 years
* Scheduled surgery
* Knee arthroscopy
* ASA Class I - III

Exclusion Criteria:

* Ipsi- or contralateral leg weakness
* Preoperative neurological deficits
* Narcotic dependent (opioid intake more than 3 months)
* Chronic pain conditions
* Significant cardiac and respiratory disease
* Coexisting hematological disorder or with deranged coagulation parameters
* Pre-existing major organ dysfunction such as hepatic and renal failure.
* Psychiatric illnesses
* Emergency surgery
* Lack of informed consent
* Allergy to any of the drugs used in the study

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the EV50 of anesthetic volume needed to produce >30% reduction of pre-injectate quadriceps strength at 20 minutes following adductor canal block. | Percentage difference before block and at 20minutes
  Measured by handheld dynamometer

SECONDARY OUTCOMES:
Reduced sensation to pin-prick around the anteromedial aspect of the knee | 20 minutes post-block
  Used to verify successful adductor canal block. scoring of either 0 - normal sensation and can feel pin-prick, 1 - touch only, 2 - no sensation of touch or pinprick
Post-operative quadriceps muscle function | Percentage difference before block and at 4 hours following block
  Measured by handheld dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- LHSC University Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Hanson NA, Derby RE, Auyong DB, Salinas FV, Delucca C, Nagy R, Yu Z, Slee AE. Ultrasound-guided adductor canal block for arthroscopic medial meniscectomy: a randomized, double-blind trial. Can J Anaesth. 2013 Sep;60(9):874-80. doi: 10.1007/s12630-013-9992-9. Epub 2013 Jul 3. PMID 23820968
- [Background] Akkaya T, Ersan O, Ozkan D, Sahiner Y, Akin M, Gumus H, Ates Y. Saphenous nerve block is an effective regional technique for post-menisectomy pain. Knee Surg Sports Traumatol Arthrosc. 2008 Sep;16(9):855-8. doi: 10.1007/s00167-008-0572-4. Epub 2008 Jun 24. PMID 18574578
- [Background] Rawal N. Postoperative pain treatment for ambulatory surgery. Best Pract Res Clin Anaesthesiol. 2007 Mar;21(1):129-48. doi: 10.1016/j.bpa.2006.11.005. PMID 17489224
- [Background] Jaeger P, Nielsen ZJ, Henningsen MH, Hilsted KL, Mathiesen O, Dahl JB. Adductor canal block versus femoral nerve block and quadriceps strength: a randomized, double-blind, placebo-controlled, crossover study in healthy volunteers. Anesthesiology. 2013 Feb;118(2):409-15. doi: 10.1097/ALN.0b013e318279fa0b. PMID 23241723
- [Background] Kim DH, Lin Y, Goytizolo EA, Kahn RL, Maalouf DB, Manohar A, Patt ML, Goon AK, Lee YY, Ma Y, Yadeau JT. Adductor canal block versus femoral nerve block for total knee arthroplasty: a prospective, randomized, controlled trial. Anesthesiology. 2014 Mar;120(3):540-50. doi: 10.1097/ALN.0000000000000119. PMID 24401769
- [Background] Muraskin SI, Conrad B, Zheng N, Morey TE, Enneking FK. Falls associated with lower-extremity-nerve blocks: a pilot investigation of mechanisms. Reg Anesth Pain Med. 2007 Jan-Feb;32(1):67-72. doi: 10.1016/j.rapm.2006.08.013. PMID 17196495
- [Background] Mayr HO, Entholzner E, Hube R, Hein W, Weig TG. Pre- versus postoperative intraarticular application of local anesthetics and opioids versus femoral nerve block in anterior cruciate ligament repair. Arch Orthop Trauma Surg. 2007 May;127(4):241-4. doi: 10.1007/s00402-006-0147-0. Epub 2006 May 23. PMID 16721618
- [Background] Chen J, Lesser JB, Hadzic A, Reiss W, Resta-Flarer F. Adductor canal block can result in motor block of the quadriceps muscle. Reg Anesth Pain Med. 2014 Mar-Apr;39(2):170-1. doi: 10.1097/AAP.0000000000000053. PMID 24553306
- [Background] Veal C, Auyong DB, Hanson NA, Allen CJ, Strodtbeck W. Delayed quadriceps weakness after continuous adductor canal block for total knee arthroplasty: a case report. Acta Anaesthesiol Scand. 2014 Mar;58(3):362-4. doi: 10.1111/aas.12244. Epub 2013 Dec 26. PMID 24372058
- [Background] Holm B, Kristensen MT, Bencke J, Husted H, Kehlet H, Bandholm T. Loss of knee-extension strength is related to knee swelling after total knee arthroplasty. Arch Phys Med Rehabil. 2010 Nov;91(11):1770-6. doi: 10.1016/j.apmr.2010.07.229. PMID 21044725
- [Background] Bohannon RW, Kindig J, Sabo G, Duni AE, Cram P. Isometric knee extension force measured using a handheld dynamometer with and without belt-stabilization. Physiother Theory Pract. 2012 Oct;28(7):562-8. doi: 10.3109/09593985.2011.640385. Epub 2011 Dec 22. PMID 22191509
- [Background] Jaeger P, Zaric D, Fomsgaard JS, Hilsted KL, Bjerregaard J, Gyrn J, Mathiesen O, Larsen TK, Dahl JB. Adductor canal block versus femoral nerve block for analgesia after total knee arthroplasty: a randomized, double-blind study. Reg Anesth Pain Med. 2013 Nov-Dec;38(6):526-32. doi: 10.1097/AAP.0000000000000015. PMID 24121608
- [Derived] Johnston DF, Sondekoppam RV, Giffin R, Litchfield R, Ganapathy S. Determination of ED50 and ED95 of 0.5% Ropivacaine in Adductor Canal Block to Produce Quadriceps Weakness: A Dose-Finding Study. Reg Anesth Pain Med. 2017 Nov/Dec;42(6):731-736. doi: 10.1097/AAP.0000000000000638. PMID 28991061